CLINICAL TRIAL: NCT05374174
Title: Validation of a Spasticity Measurement Tool
Status: Active, not recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Director Single Motor Unit Laboratory, Shirley Ryan AbilityLab
Other Study IDs: STU00216437
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Spasticity; Hyperreflexia; Clonus; Hypertonia
MeSH Terms: conditions — Stroke; Muscle Spasticity; Reflex, Abnormal; Muscle Hypertonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement Group: All participants will have their arm spasticity to be measured using standard clinical scales
  Interventions: Diagnostic Test: Tardieu Scale for Spasticity

INTERVENTIONS:
Diagnostic Test: Tardieu Scale for Spasticity — The clinician will rotate the elbow joint at various speeds while the participant sits relaxed.

SUMMARY:
The objective of this project is to investigate the validity of a handheld spasticity measurement tool against standard clinical measurements of spasticity. We propose the testing apparatus will accurately provide an equivalent clinical measure of spasticity while also providing a more precise estimation of spastic response in persons with stroke.

DETAILED DESCRIPTION:
An ongoing conversation amongst clinicians exists on how to properly define, measure, and manage spasticity. The standard measurement tools are the Modified Ashworth Scale (MAS) and the Tardieu scale, although both of these lack reliability and specificity, causing variability between clinicians and a lack of accurate spasticity measurement. In addition, some have concerns about whether the MAS measures true spasticity at all. Due to this lack of trust in these scales, clinicians often use them as a communication tool to identify the presence of spasticity, rather than as reliable quantifiable outcome measurements.

The MAS and Tardieu function mainly on the principal of catch, a limb is moved slowly by a clinician through the available range of motion, and then quickly. Hyperactive muscles are sensitive to velocity dependent stretch and will activate a reflex if quickly perturbed. In both the MAS and Tardieu, the catch location is noted and translated into a score. In MAS the catch location is only noted in three distinct ranges; with the Tardieu Scale the catch angle is remembered by the clinician and recorded after the movement with a standard goniometer.

Here we will test a new handheld spasticity measurement tool MITSS (Modified Intelligent Tardieu Scale for Spasticity), which is essentially a 3-DOF digital goniometer, to quantify the catch angle as well as general forces at the joint.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Able to provide informed consent
* History of unilateral stroke

Exclusion Criteria:

* Orthopedic injuries or surgeries that would impact arm function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who have experienced a unilateral stroke
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Catch angle | Baseline
  Elbow angle in which there is a marked increase in tone while rotating quickly. This is measured while the clinician is wearing the MITSS and rotating participant's elbow slowly and quickly through the range of motion. This measure will be taken at 2 minute increments over 30 minutes

SECONDARY OUTCOMES:
Modified ashworth score | Baseline
  Clinical measure of tone in the elbow. Participant is relaxed while the clinician rotates the elbow through the range of motion. Scale is rated from 0-4 where 0 is tone, 1 is slight increase in tone, catch at end of range of motion, 1+ is slight increase in tone, catch in 1st half of range of motion, 2 is increased tone throughout range of motion, but still moveable, 3 is a considerable increase in tone, and 4 is a rigid limb. This measure will be taken at 2 minute increments over 30 minutes
Tardieu Spasticity Score | Baseline
  Clinical measure of catch angle during fast elbow rotation. Participant is relaxed while the clinician rotates the elbow through the range of motion quickly and slowly. Angle of catch is recorded for this scale, measured with goniometer. The quantitative score is from 0-4, It is scored as 0, no resistance, 1 slight resistance, 2 clear catch followed by release, 3 clonus which dissipates in less than 10 seconds, and 4 is clonus lasting more than 10 seconds. This measure will be taken at 2 minute increments over 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: William Z Rymer, MD, PhD, Principal Investigator — Director, Single Motor Unit Laboratory
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided